CLINICAL TRIAL: NCT03665688
Title: Induction of Labor in Women With Unfavorable Cervix: Randomized Controlled Trial Comparing Outpatient to Inpatient Cervical Ripening Using Dilapan-S® (HOMECARE)
Brief Title: Comparing Outpatient to Inpatient Cervical Ripening Using Dilapan-S®
Acronym: HOMECARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: Medicem International CR s.r.o. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18-0132
Record Dates: First submitted 2018-08-30; First posted 2018-09-11 (Actual); Results first posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Labor, Induced; Cervix Uteri-Diseases
Keywords: Cervical ripening; Labor induction; Outpatient; Mechanical; Hygroscopic

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Outpatient Dilapan-S (Experimental): After Dilapan-S® placement, subjects will be given the option to either return home or to stay in a hotel if transportation is an issue.
  Subjects will also be instructed to return to L&D unit 12 hours after insertion, or earlier if any excessive bleeding, rupture of membranes, pain or other concerns (contractions, decreased fetal movement) develop before the 12 hours
  Interventions: Device: Outpatient Dilapan-S
- Inpatient Dilapan-S (Active Comparator): After Dilapan-S® placement, subjects will be admitted to L&D unit and standard clinical protocol will be initiated for cervical ripening and labor induction. During the period of 12 hours of cervical ripening subject is to remain "nothing per os" (NPO), "nothing per vagina" and undergo continuous fetal heart rate monitoring. No other interventions are to occur during this period of 12 hours, unless clinically indicated.
  Interventions: Device: Inpatient Dilapan-S

INTERVENTIONS:
Device: Outpatient Dilapan-S — After Dilapan-S placement, subjects will be given the option to either return home or to stay in a hotel if transportation is an issue. Subjects will also be instructed to return to L&D unit 12 hours after insertion, or earlier if any excessive bleeding, rupture of membranes, pain or other concerns (contractions, decreased fetal movement) develop before the 12 hours. After the designated 12 hours' time or earlier, if indicated, subjects are to return and to be admitted to L&D unit for standard protocol of labor induction.
  Other Names: Outpatient cervical ripening with Dilapan-S
  Arms: Outpatient Dilapan-S
Device: Inpatient Dilapan-S — After Dilapan-S placement, subjects will be admitted to L&D unit and standard clinical protocol will be initiated for cervical ripening and labor induction. During the period of 12 hours of cervical ripening subject is to remain "nothing per os" (NPO), "nothing per vagina" and undergo continuous fetal heart rate monitoring. No other interventions are to occur during this period of 12 hours, unless clinically indicated.
  Other Names: Inpatient cervical ripening with Dilapan-S
  Arms: Inpatient Dilapan-S

SUMMARY:
The target population for our study is women who present for induction of labor. If there is a decision by the obstetrical team to place a mechanical dilator for cervical ripening, the obstetrical team will notify the research staff so that the patient may be screened for the study. If the subject is eligible for the trial, written informed consent will be obtained by person-to-person contact. The PI, study coordinator, or a collaborator will be responsible for the informed consent procedure. After informed consent is obtained and Dilapan-S is placed, the patient will be randomized to the Outpatient or the Inpatient group.

DETAILED DESCRIPTION:
Group Assigned to Outpatient Cervical Ripening After Dilapan-S® placement, subject will be monitored for at least 30 minutes. If no contraindications, such as tachysystole, active vaginal bleeding, rupture of membranes or nonreassuring fetal testing (defined as minimal or absent variability, abnormal baseline, or presence of decelerations) evidence of labor, or other serious medical conditions deemed by the clinical staff or the attending physician to preclude outpatient cervical ripening develop after insertion, the subjects will be randomized. After randomization subject will record the pain she experienced during insertion in the patient's survey (see Appendix 3). Those subjects randomized to outpatient ripening will be given the option to either return home or to stay in a hotel if transportation is an issue. The cost for the hotel will be covered by the study budget. Subjects will be allowed to ambulate, shower and perform regular activity during that period. "Nothing per vagina" will be allowed (incl. intercourse, tampons etc.).

Group Assigned to Inpatient Cervical Ripening Subjects randomized to inpatient management will be admitted to L&D unit and standard clinical protocol will be initiated for cervical ripening and labor induction. During the period of 12 hours of cervical ripening subject is to remain "nothing per os" (NPO), "nothing per vagina" and undergo continuous fetal heart rate monitoring. No other interventions are to occur during this period of 12 hours, unless clinically indicated.

Labor Induction and Labor Management of the subject after the initial 12 hours of pre-induction or following the earlier removal or spontaneous expulsion of the dilator will be the same for both groups and at the discretion of the clinical team. Additional ripening (mechanical or prostaglandins) and/or oxytocin may or may not be needed. If needed, duration, type and dose of additional ripening agents and oxytocin will be documented.

Routine intrapartum care will be provided and relevant data collected by the subject's managing obstetrical team.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant woman whose plan of care is induction of labor
2. Maternal age between 18 and 45 years
3. Understanding and capable to sign informed consent
4. Singleton pregnancy
5. Gestational age ≥ 37 0/7 weeks (based on a sure last menstrual period or a first trimester dating ultrasound)
6. Live fetus in cephalic presentation
7. Intact membranes
8. Pelvic exam (sterile vaginal exam) of less than or equal to 3cm and at most 60% effaced

Exclusion Criteria:

1. Active labor
2. Active genital herpes
3. Chorioamnionitis
4. Transfundal uterine or cervical surgery
5. Previous cesarean delivery
6. Non-reassuring fetal status
7. Need for continuous maternal or fetal monitoring during ripening
8. Contraindication for vaginal delivery
9. Active vaginal bleeding
10. Abnormal placental location or adherence (placenta previa or unresolved low lying placenta)
11. Estimated fetal weight > 5000 g (non diabetic) or > 4500 g (diabetic)
12. Intrauterine growth restriction (estimated fetal weight <10 percentile)
13. Oligohydramnios (amniotic fluid index < 5cm or deep vertical pocket of < 2 cm)
14. Fetal anomaly
15. Need for inpatient care (e.g. hypertension, insulin-dependent diabetes)
16. Poor or no access to a telephone and cannot be placed in the hotel
17. Absence of support person ( no adult accompanying the subject during outpatient cervical ripening period)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 338 (Actual)
Dates: Start 2018-11-07 (Actual); Primary Completion 2021-11-05 (Actual); Study Completion 2021-11-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Saad, MD, Principal Investigator — The University of Texas Medical Branch, Galveston
Locations (2):
- United States (2):
  - Columbia University Irving Medical Center, New York, New York
  - UTMB Galveston, Galveston, Texas

REFERENCES:
- [Background] Thiery M, De Boever J, Merchiers E, Martens G. Hormones and cervical ripening. Am J Obstet Gynecol. 1989 May;160(5 Pt 1):1251-3. doi: 10.1016/0002-9378(89)90207-x. No abstract available. PMID 2524974
- [Background] Grobman WA, Rice MM, Reddy UM, Tita ATN, Silver RM, Mallett G, Hill K, Thom EA, El-Sayed YY, Perez-Delboy A, Rouse DJ, Saade GR, Boggess KA, Chauhan SP, Iams JD, Chien EK, Casey BM, Gibbs RS, Srinivas SK, Swamy GK, Simhan HN, Macones GA; Eunice Kennedy Shriver National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. Labor Induction versus Expectant Management in Low-Risk Nulliparous Women. N Engl J Med. 2018 Aug 9;379(6):513-523. doi: 10.1056/NEJMoa1800566. PMID 30089070
- [Background] Wilkinson C, Adelson P, Turnbull D. A comparison of inpatient with outpatient balloon catheter cervical ripening: a pilot randomized controlled trial. BMC Pregnancy Childbirth. 2015 May 28;15:126. doi: 10.1186/s12884-015-0550-z. PMID 26018581
- [Background] Wilkinson C, Bryce R, Adelson P, Turnbull D. A randomised controlled trial of outpatient compared with inpatient cervical ripening with prostaglandin E(2) (OPRA study). BJOG. 2015 Jan;122(1):94-104. doi: 10.1111/1471-0528.12846. Epub 2014 May 14. PMID 24824157
- [Background] Henry A, Madan A, Reid R, Tracy SK, Austin K, Welsh A, Challis D. Outpatient Foley catheter versus inpatient prostaglandin E2 gel for induction of labour: a randomised trial. BMC Pregnancy Childbirth. 2013 Jan 29;13:25. doi: 10.1186/1471-2393-13-25. PMID 23356673
- [Background] Kruit H, Heikinheimo O, Ulander VM, Aitokallio-Tallberg A, Nupponen I, Paavonen J, Rahkonen L. Foley catheter induction of labor as an outpatient procedure. J Perinatol. 2016 Aug;36(8):618-22. doi: 10.1038/jp.2016.62. Epub 2016 Apr 14. PMID 27078202
- [Background] Sciscione AC, Muench M, Pollock M, Jenkins TM, Tildon-Burton J, Colmorgen GH. Transcervical Foley catheter for preinduction cervical ripening in an outpatient versus inpatient setting. Obstet Gynecol. 2001 Nov;98(5 Pt 1):751-6. doi: 10.1016/s0029-7844(01)01579-4. PMID 11704164
- [Background] Diederen M, Gommers J, Wilkinson C, Turnbull D, Mol B. Safety of the balloon catheter for cervical ripening in outpatient care: complications during the period from insertion to expulsion of a balloon catheter in the process of labour induction: a systematic review. BJOG. 2018 Aug;125(9):1086-1095. doi: 10.1111/1471-0528.15047. Epub 2018 Jan 10. PMID 29211328
- [Background] Gupta J, Chodankar R, Baev O, Bahlmann F, Brega E, Gala A, Hellmeyer L, Hruban L, Maier J, Mehta P, Murthy A, Ritter M, Saad A, Shmakov R, Suneja A, Zahumensky J, Gdovinova D. Synthetic osmotic dilators in the induction of labour-An international multicentre observational study. Eur J Obstet Gynecol Reprod Biol. 2018 Oct;229:70-75. doi: 10.1016/j.ejogrb.2018.08.004. Epub 2018 Aug 3. PMID 30107363
- [Background] Kuper SG, Jauk VC, George DM, Edwards RK, Szychowski JM, Mazzoni SE, Wang MJ, Files P, Tita AT, Subramaniam A, Harper LM. Outpatient Foley Catheter for Induction of Labor in Parous Women: A Randomized Controlled Trial. Obstet Gynecol. 2018 Jul;132(1):94-101. doi: 10.1097/AOG.0000000000002678. PMID 29889751
- [Derived] Saad AF, Gavara R, Senguttuvan RN, Goncharov AD, Berry M, Eid J, Goldman B, Nutter A, Moutos CP, Wang AM, Saade GR. Outpatient Compared With Inpatient Preinduction Cervical Ripening Using a Synthetic Osmotic Dilator: A Randomized Clinical Trial. Obstet Gynecol. 2022 Oct 1;140(4):584-590. doi: 10.1097/AOG.0000000000004942. Epub 2022 Sep 7. PMID 36083097
- [Derived] Alfirevic Z, Gyte GM, Nogueira Pileggi V, Plachcinski R, Osoti AO, Finucane EM. Home versus inpatient induction of labour for improving birth outcomes. Cochrane Database Syst Rev. 2020 Aug 27;8(8):CD007372. doi: 10.1002/14651858.CD007372.pub4. PMID 32852803

RESULTS

PARTICIPANT FLOW:
Groups:
- Outpatient Dilapan-S: After Dilapan-S® placement, subjects will be given the option to either return home or to stay in a hotel if transportation is an issue.
  Subjects will also be instructed to return to L&D unit 12 hours after insertion, or earlier if any excessive bleeding, rupture of membranes, pain or other concerns (contractions, decreased fetal movement) develop before the 12 hours
  Outpatient Dilapan-S: After Dilapan-S placement, subjects will be given the option to either return home or to stay in a hotel if transportation is an issue. Subjects will also be instructed to return to L&D unit 12 hours after insertion, or earlier if any excessive bleeding, rupture of membranes, pain or other concerns (contractions, decreased fetal movement) develop before the 12 hours. After the designated 12 hours' time or earlier, if indicated, subjects are to return and to be admitted to L&D unit for standard protocol of labor induction.
Period: Overall Study
Arm/Group | Outpatient Dilapan-S | Inpatient Dilapan-S
Started | 167 | 171
Completed | 167 | 171
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Outpatient Dilapan-S | Inpatient Dilapan-S | Total
Number analyzed (Participants) | 167 | 171 | 338
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.2 (5.6) | 25.9 (5.6) | 25.5 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 167 | 171 | 338
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 120 | 112 | 232
  Not Hispanic or Latino | 47 | 59 | 106
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 167 | 171 | 338

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Hospital Stay Longer Than 48 Hours
Description: Rate of hospital stay longer than 48 hours (from admission to discharge)
Time Frame: 72 hours or discharge home time, whichever occurs first
Measure: Count of Participants; unit: Participants
Arm/Group | Outpatient Dilapan-S | Inpatient Dilapan-S
Number analyzed (Participants) | 167 | 171
Participants | 89 | 152

2. Secondary Outcome: Number of Participants With Vaginal Deliveries 2-4 Days
Description: Rate of vaginal deliveries (%)
Time Frame: 2-4 days
Measure: Count of Participants; unit: Participants
Arm/Group | Outpatient Dilapan-S | Inpatient Dilapan-S
Number analyzed (Participants) | 167 | 171
Participants | 125 | 128

3. Secondary Outcome: Number of Participants With Vaginal Deliveries - 24 Hours
Description: Rate of vaginal deliveries within 24 hours since admission to hospital (%)
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Outpatient Dilapan-S | Inpatient Dilapan-S
Number analyzed (Participants) | 167 | 171
Participants | 117 | 86

4. Secondary Outcome: Time From Hospital Admission to Active Stage of Labor
Description: Time from hospital admission to reach active stage of labor defined as cervical dilation of ≥ 6 cm (in minutes)
Time Frame: 1-2 days
Measure: Median (Full Range); unit: minutes
Arm/Group | Outpatient Dilapan-S | Inpatient Dilapan-S
Number analyzed (Participants) | 167 | 171
minutes | 545 [492 to 690] | 1183 [1141 to 1265]

5. Secondary Outcome: Change in Bishop Score From Insertion of Device to Extraction
Description: Change in Bishop score (based on cervical dilation, position of cervix, effacement of cervix, fetal station and softness of cervix) . Calculated as Bishop score value at 12 hours minus value at baseline. Bishop score ranges from zero to 13, with zero meaning you're not ready for induction and 13 indicating a better chance for successful induction. A higher score means that labor is closer, and that induction has a good chance of being successful.
Time Frame: 12 hours
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Outpatient Dilapan-S | Inpatient Dilapan-S
Number analyzed (Participants) | 167 | 171
score on a scale | 2 [1 to 4] | 2 [1 to 4]

6. Secondary Outcome: Number of Participants With Operative Vaginal Delivery
Description: Rate of operative vaginal deliveries (%)
Time Frame: 1-4 days
Measure: Count of Participants; unit: Participants
Arm/Group | Outpatient Dilapan-S | Inpatient Dilapan-S
Number analyzed (Participants) | 167 | 171
Participants | 6 | 5

7. Secondary Outcome: Number of Participants With Cesarean Delivery
Description: Rate of caesarean deliveries (%)
Time Frame: 1-4 days
Measure: Count of Participants; unit: Participants
Arm/Group | Outpatient Dilapan-S | Inpatient Dilapan-S
Number analyzed (Participants) | 167 | 171
Participants | 42 | 43

ADVERSE EVENTS:
Time Frame: at the time the participant are enrolled into the study, up to 3 years
Arm/Group | Outpatient Dilapan-S | Inpatient Dilapan-S
All-Cause Mortality (participants affected / at risk) | 0/167 | 0/171
Serious Adverse Events (participants affected / at risk) | 0/167 | 0/171
Other Adverse Events (participants affected / at risk) | 0/167 | 0/171

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-19): https://cdn.clinicaltrials.gov/large-docs/88/NCT03665688/Prot_SAP_002.pdf